CLINICAL TRIAL: NCT07297108
Title: Study of the Survival and Success of Endodontic Posts Exclusively Using the CAD/CAM Digital Method After 5 Years of Intraoral Use
Brief Title: Endodontic Posts Using the CAD/CAM Digital Method.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Petros Mourouzis, Assistant Professor, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 203/30-11-2023
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Endodontic Treatment; Tooth Restoration
Keywords: CAD/CAM; intraoral Scanners; post fabrication; endodontic posts

STUDY DESIGN:
Intervention Model Description: This study uses a parallel-group interventional model in which patients are allocated to different treatment arms corresponding to distinct types of indirect restorations or restorative materials. Each participant receives only the assigned intervention, performed under standardized preparation, adhesive, and cementation protocols. The model allows comparison of clinical performance, survival, and success rates among the different restorative approaches. All groups are followed longitudinally using predefined clinical and radiographic criteria to assess restoration integrity, functional stability, biological compatibility, and the need for repair or replacement.
Masking Description: This is an open-label trial; no parties are masked in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Lithium Disilicate CAD/CAM Posts (Experimental): Patients in this arm receive custom CAD/CAM posts fabricated from lithium disilicate. All posts are designed, milled, and cemented using standardized preparation, adhesive, and cementation protocols. Clinical follow-up evaluates post survival, success rates, biological response, and the need for repair or replacement over time.
  Interventions: Device: Lithium Disilicate CAD/CAM Post
- Active Comparator: Polymer-Based CAD/CAM Posts (Active Comparator): Patients in this arm receive custom CAD/CAM posts fabricated from high-performance polymer materials. Posts are manufactured and cemented using the same standardized clinical workflow applied in Arm 1. This arm allows comparison of survival, success rates, functional stability, and biological outcomes relative to lithium disilicate CAD/CAM posts.
  Interventions: Device: Active Comparator: Polymer-Based CAD/CAM Posts

INTERVENTIONS:
Device: Lithium Disilicate CAD/CAM Post — Patients in this arm receive custom CAD/CAM posts fabricated from lithium disilicate. All posts are designed, milled, and cemented using standardized preparation, adhesive, and cementation protocols. Clinical follow-up evaluates post survival, success rates, biological response, and the need for repair or replacement over time.
  Arms: Experimental: Lithium Disilicate CAD/CAM Posts
Device: Active Comparator: Polymer-Based CAD/CAM Posts — Patients in this arm receive custom CAD/CAM posts fabricated from high-performance polymer materials. Posts are manufactured and cemented using the same standardized clinical workflow applied in Arm 1. This arm allows comparison of survival, success rates, functional stability, and biological outcomes relative to lithium disilicate CAD/CAM posts.
  Arms: Active Comparator: Polymer-Based CAD/CAM Posts

SUMMARY:
This study investigates the survival and success rates of endodontic posts exclusively fabricated using the CAD/CAM digital method over a period of 5 years of intraoral use. The objective is to evaluate the efficacy and long-term outcomes of the digital approach compared to traditional techniques, aiming to determine the reliability and precision of CAD/CAM technology in the fabrication of endodontic post restorations.

DETAILED DESCRIPTION:
This clinical study aims to evaluate the survival and success rates of endodontic posts exclusively fabricated using the CAD/CAM digital method over a period of 5 years of intraoral use. The study focuses on the utilization of advanced digital technology for the design and fabrication of endodontic posts, which replaces traditional impression-taking and analog methods.

Participants in the study will undergo treatment where digital intraoral scanners will capture the post-space anatomy, and CAD software will be used to design custom posts that are then milled using CAM technology. The fabricated posts will be evaluated for fit, stability, and clinical performance over a prolonged period.

The primary outcome measures include the survival rate of the posts (absence of dislodgement or failure) and the success rate, which incorporates the functional and aesthetic integration of the post with the surrounding dental structures. Secondary outcomes will assess the incidence of complications such as root fractures, debonding, and endodontic failure.

This study distinguishes itself by exclusively using the digital CAD/CAM approach, with no involvement of traditional methods, ensuring precision and consistency in post fabrication. It aims to provide comprehensive data on the effectiveness and reliability of CAD/CAM technology for endodontic applications, offering insights that could influence clinical protocols and materials used in restorative dentistry

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 to 70 years
* Patients requiring endodontic treatment with post placement
* Individuals with adequate tooth structure to support a post restoration
* Patients who consent to participate and commit to follow-up visits for a period of 5 years
* Good overall oral health with no active periodontal disease

Exclusion Criteria:

* Patients with systemic conditions that could affect oral health or healing (e.g., uncontrolled diabetes or immune-compromising diseases)
* Individuals with severe periodontal disease or compromised tooth structure unsuitable for post placement
* Pregnant or breastfeeding women
* Patients unwilling or unable to commit to the 5-year follow-up period
* Individuals with allergies or adverse reactions to dental materials used in the CAD/CAM process
* Minimum Age = 18 Years and Maximum Age = 70 Years

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Survival Rate of CAD/CAM Endodontic Posts | Assessed over a period of 5 years post-placement
  The primary outcome measure is the survival rate of endodontic posts fabricated using the CAD/CAM digital method. Survival is defined as the post remaining in situ without any signs of dislodgement, root fracture, or clinical failure necessitating replacement. Posts will be evaluated periodically to monitor their clinical performance and integrity, ensuring that no adverse events such as post loosening or tooth failure occur

CONTACTS AND LOCATIONS:
Overall Officials: Kosmas Tolidis, Professor, Study Chair — School of Dentistry, Aristotle University of Thessaloniki
Locations (1):
- School of Dentisty, Aristotle University of Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) from this study will not be shared due to privacy and confidentiality concerns. The data collected includes sensitive patient information, and sharing it publicly may compromise participant anonymity and violate ethical guidelines. Furthermore, the study does not have the necessary infrastructure in place to ensure secure and compliant sharing of IPD with other researchers.